CLINICAL TRIAL: NCT05546710
Title: Post-market Clinical Investigation of High-Volume Anesthesia (Local Tumescent Anesthesia) Used With the miraDry Treatment for Axillary Hyperhidrosis
Brief Title: miraDry Post Market Tumescent Anesthesia Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision to pivot priorities
Sponsor: miraDry, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0024
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Hyperhidrosis; Axillary Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, open-label, multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): miraDry treatment
  Interventions: Device: miraDry treatment

INTERVENTIONS:
Device: miraDry treatment — The miraDry device is non-invasive and uses microwave energy, focused at the dermal/hypodermal interface, to thermally impact the sweat glands. The treatment area is identified (hair bearing area of the axilla) and high-volume anesthesia is delivered. The miraDry template is selected based upon the size of the treatment area and temporarily applied to the patient's skin. A new miraDry bioTip is attached to the miraDry Handpiece for each treatment session. The Handpiece is then placed on the surface of the skin in the area to be treated. The treatment cycle is activated by a button on the Handpiece. Multiple placements of the Handpiece are required to treat a full axilla in one treatment session.
  Other Names: Tumescent Anesthesia (high-volume anesthesia)

SUMMARY:
This clinical trial will collect data on the safety and efficacy of the miraDry treatment when High Volume Anesthesia (Tumescent Anesthesia) is used as an alternate method of anesthetizing the axilla prior to the miraDry System being used. MiraDry system was FDA cleared in 2011 for the treatment of primary axillary hyperhidrosis. The miraDry system is also CE-marked.

DETAILED DESCRIPTION:
Hyperhidrosis is a condition defined as sweating beyond what is physiologically required by the body (excessive sweating). Hyperhidrosis sufferers have been shown to suffer from anxiety, social and occupational impairment and limitation of exercise, recreation, and leisure. In addition to psychological and social issues, hyperhidrosis sufferers see significant financial burden from their condition. The costs of treatments which need to be repeated chronically and replacing clothing which is permanently stained and unwearable can amount to significant expenditures over time.

Many physicians using the miraDry System are using alternative methods for anesthetizing the axilla; the most common is infiltrative local tumescent anesthesia (LTA) at a high volume. miraDry often calls this method as High Volume Anesthesia (HVA) and the two terms are used interchangably. Tumescent anesthesia is commonly used for various dermatologic surgery procedures. This method involves using a larger volume of fluid with a lower concentration of lidocaine; the fluid is introduced under the skin through a few small injection sites and infiltrated into the desired region. For this application using the tumescent technique, between 100 and 300 cc's of fluid per axilla would be introduced subcutaneously, depending on the size of the axilla.

This clinical trial will collect data on the safety and efficacy when High Volume Anesthesia is used as an alternate method of anesthetizing the axilla prior to the miraDry System being used. The investigators participating in this study are experts in the administration of tumescent anesthesia for dermatologic applications.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (aged ≥18 years) at time of consent.
2. A HDSS score of 3 or 4.
3. Excess sweating evidenced by at least two of the following:

a. Impairs daily activities b. Frequency of at least one episode per week c. Age of onset less than 25 years old d. Positive family history e. Cessation of focal sweating during sleep d) In the opinion of the physician, treatment with the miraDry System is technically feasible and clinically indicated.

e) Willing and able to comply with protocol requirements and all study visits. f) Female patients of child-bearing potential must not be pregnant or lactating and must agree to not become pregnant during the course of the study.

Exclusion Criteria:

1. A cardiac pacemaker or cardiac defibrillator or other electronic implant.
2. Requires supplemental oxygen.
3. Known resistance to or history of intolerance of local anesthesia including lidocaine and epinephrine.
4. Secondary excess sweating due to medications, infections, malignancy.
5. Evidence of active infection or prone to infection.
6. Prior liposuction or other dissection surgery for axillary excess sweating.
7. Oral anticholinergic medication use (e.g., Glycopyrrolate) or cholinomimetic medication use within the last 4 weeks or planned use during the study's follow-up phase.
8. Taking any other medication that may hinder post-procedure recovery and/or healing.
9. Botulinum treatment of the axilla within the last 12 months.
10. Currently participating in or recently participated in another clinical trial (within the last 30 days).
11. History of or current neurologic deficit in the treatment area and/or limb.
12. History of cancer with the exception of (1) successfully treated basal cell or squamous cell carcinoma of the skin or (2) a history of successfully treated cancer that have been disease-free for five years.
13. Any history of cysts, hidradenitis suppurativa, etc.
14. Pre-existing conditions at the time of enrollment that overlap with the list of anticipated AEs (Section 6.1).
15. Prior treatment in axillary area with miraDry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of device and/or treatment related serious adverse events (SAEs) | 30 days
  Incidence of device and/or treatment related serious adverse events (SAEs)
Responder rate: defined as a study participant that reports a Hyperhidrosis Severity Scale (HDSS) score of 1 or 2 | 30 days
  Responder rate: defined as a study participant that reports a Hyperhidrosis Severity Scale (HDSS) score of 1 or 2

SECONDARY OUTCOMES:
Incidence of device and/or treatment related SAEs and AEs | 6 months
  Incidence of device and/or treatment related SAEs and AEs
Responder rate: HDSS score of 1 or 2 | 3 and 6 months
  Responder rate: HDSS score of 1 or 2
Change in Quality of Life from baseline as measured by the Dermatology Life Quality Index (DLQI) | 30 days, 3 months, and 6 months
  Change in Quality of Life from baseline as measured by the Dermatology Life Quality Index (DLQI)
Change in odor assessment score from baseline | 30 days, 3 months, and 6 months
  Change in odor assessment score from baseline